CLINICAL TRIAL: NCT03075189
Title: Increased Focus on Protein Intake Among Geriatric Patients During Hospitalization: Serving and Acceptance of Protein Enriched Meals in the Morning and Before Bedtime, as Well as Nutritional Guidance by a Clinical Dietician.
Brief Title: Increased Focus on Protein Intake Among Geriatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Slagelse Hospital (Other); Arla Foods (Industry)
Responsible Party: Principal Investigator, Lars Holm, Associate professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16045350
Record Dates: First submitted 2017-02-10; First posted 2017-03-09 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Geriatric Diseases
Keywords: Frailty; geriatric; hospitalized; enrichment; whey protein; protein intake; sarcopenia; dietary counseling
MeSH Terms: conditions — Frailty; Sarcopenia

STUDY DESIGN:
Intervention Model Description: Inclusion and testing of intervention and control group is carried out at the same time
Who Masked: Investigator, Outcomes Assessor
Masking Description: Two of the study officials will be masked and therefore responsible for testing the participants at baseline, at discharge and follow-up - and in charge of data processing.
  Contrary to the masked officials two non-masked officials are responsible for randomization, serving of meals, diet registration and dietary counseling.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein supplement (Experimental): During hospitalization the intervention group will receive a protein enriched snack/meal in the morning and before bedtime. They will be given 15 gr of protein every morning, and the meal before bedtime will vary in protein content according to the individual needs. Diet registration will be carried out every day during hospitalization. At discharge, participants in the intervention will be instructed and advised with focus on consuming more protein at home.
  Diet registration and testing at baseline, discharge and follow-up.
  Interventions: Dietary Supplement: Whey protein supplement
- Standard treatment (No Intervention): The control group are having the ordinary hospital diet and are following normal guidelines. They are not offered the protein focused counseling at discharge.
  Diet registration and testing at baseline, discharge and follow-up.

INTERVENTIONS:
Dietary Supplement: Whey protein supplement — During hospitalization the intervention group will receive a whey protein enriched snack/meal in the morning and before bedtime. They will be given 15 gr of protein every morning, and the meal before bedtime will vary in protein content according to the individual needs. Diet registration will be carried out every day during hospitalization. At discharge, participants in the intervention will be instructed and advised with focus on consuming more protein at home.
  The control group are having the ordinary hospital diet and are following normal guidelines. They are not offered the protein focused counseling at discharge.
  Both groups have diet registration and testing at baseline, discharge and follow-up.
  Arms: Protein supplement

SUMMARY:
Up to approximately 38 (unknown drop-out rate) geriatric patients (at least 65 years old) are recruited from a Geriatric ward at Slagelse Sygehus. After inclusion and baseline measurements, each individual will be randomized into either an intervention or control group arranged in blocks of 8 The intervention group (n≤19) will receive protein enriched snacks/dishes in the morning and late evening, before bedtime. Moreover, upon discharge the intervention group will receive individual dietary counseling focusing on choosing protein-rich foods and on protein rich meals. The control group (n≤19) will receive normal hospital food without enrichment and no dietary counseling at discharge. In both groups the following data will be obtained: recorded protein intake, anthropometric measurements (weight, height, body composition estimated with bioimpedance), functional ability (De Morton Mobility Index (DEMMI) and Barthels ADL-index), hand grip strength, sarkopenic status (SARC-F), quality of life (EQ-5D-3L), length of stay (LOS) and readmissions (within 30 days after discharge). During hospitalization food intake will be registered, as well as 24 hour recall interviews and food frequency questionnaires will be done at follow-up visits.

Assessments will be performed at baseline, on the day of discharge and 4 weeks after discharge (follow up).

The primary outcome is change in protein intake from Baseline to 4 weeks after discharge.

The hypothesis is that serving of individually selected protein enriched snack/dish in the morning and before bedtime during hospitalization results in higher protein intake during hospitalization and that this experience combined with dietary counseling at discharge, results in a higher protein intake at 28 days after discharge. Further, we hypothesize that the increased protein intake will affect functional level, hand grip strength, sarcopenic status and quality of life in geriatric patients and will lead to shorter LOS and fewer readmission frequency.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥65 år and admitted to the geriatric ward at Slagelse Hospital.
* Expected length-of-stay, LOS: more than 3 days
* Normal kidney function. (As long as the kidney values remain stable during the intervention it is deemed safe to take part, as the amount of protein given will not exceed the amount recommended by the Danish authorities.

Exclusion Criteria:

* Dysphagia
* Patients exclusively fed by tube/probe or parenteral nutrition.
* Gastrointestinal problems, that makes normal food intake impossible.
* People suffering from dementia, deliriousness or severe memory loss
* Patients abusing alcohol
* Patients in isolation
* Terminal patients
* Patients that do not speak Danish or English
* Patients suffering from food allergies/intolerances that makes it impossible to accommodate to the protein enriched foods.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Protein intake | Change from baseline up to 6 weeks
  Dietary recordings with focus on protein intake are collected during hospitalization and at follow up. The total intake of protein per day is assessed.

SECONDARY OUTCOMES:
Change in grib strength | Baseline, up to 8 days, up to 6 weeks
  Isometric hand grib strength. The patients sit in an upright position, resting their arm and holding a hand dynamometer in the non-dominant arm. Then a maximum pressure test is performed with the hand and the strength is recorded.
De Morton Mobility Index (DEMMI) | Baseline, up to 8 days, up to 6 weeks
  A mobility test used as standard procedure when admitted to the geriatric ward. The test contains 15 tasks of different difficulty, such as rising from a chair, static and dynamic balance and walk.
Barthel ADL-index | Baseline, up to 8 days, up to 6 weeks
  Testing the patient's ability to perform different activities of daily living, such as eating, movement, personal hygiene and toilet visits. The test consists of 10 steps, and each step results in a score from 5-15 when performed by the patient.
SARC-F | Baseline, up to 8 days, up to 6 weeks
  A screening tool, where the patient is asked about different physical parameters in relation to the risk of developing sarcopenia: parameters such as falls, assistance to walk, general strength, rise from a chair and walk on stairs.
EQ-5D-3L | Baseline, up to 8 days, up to 6 weeks
  A questionnaire focusing on self-perceived quality of life. The questions are divided into 5 categories: mobility, personal hygiene, pain, anxiety and ability to perform ADL-activities.
Length of stay (LOS) | Up to 8 days (after baseline)
  Based on information from electronic patient journal. LOS is defined from day of admission to day of discharge.
Readmission | Up to 6 weeks (after baseline)
  Based on information from electronic patient journal and is defined as a readmission less than 30 days after discharge.
Anthropometric measures | Change from baseline up to 6 weeks
  Weight is measured to make individual calculations of protein and energy needs.
Bioimpedance | Up to 2 days and up to 6 weeks
  Measurement of fat and muscle distribution in the body. Is measured on day 2-3 after inclusion because of possible irregularities in fluid balance at admission to the hospital and after surgery
24h recall interview | Up to 6 weeks
  Interviewers asks the participant about their dietary intake through the last 24 hours. A standard technique with four steps is used for this interview.
Food frequency questionnaire | Up to 6 weeks
  A list containing the most protein rich food items are given to the participant and they are asked how frequent they have had the items during the last 4 weeks after discharge.
Nutrition related complications | Up to 8 days and up to 6 weeks.
  Infections, falls and decreased wound healing

CONTACTS AND LOCATIONS:
Locations (1):
- Slagelse Hospital, Slagelse, Ingemannsvej 18, Denmark

IPD SHARING:
Plan to Share IPD: No